CLINICAL TRIAL: NCT02797847
Title: A Phase 1, Randomized, Single-Blind, Placebo Controlled, Single-Ascending Dose, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics Study of Subcutaneously Administered ALN-TTRSC02 in Healthy Subjects
Brief Title: A Safety and Tolerability Study of an Investigational Drug, ALN-TTRSC02, in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALN-TTRSC02-001; 2015-005803-98 (EudraCT Number)
Record Dates: First submitted 2016-05-18; First posted 2016-06-14 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Transthyretin-mediated Amyloidosis (ATTR Amyloidosis)
Keywords: TTR-mediated Amyloidosis; Amyloidosis, Hereditary; Amyloid Neuropathies, Familial; Familial Amyloid Polyneuropathies; Amyloid Neuropathies; Amyloidosis, Hereditary, Transthyretin-Related; Familial Amyloidosis; RNAi therapeutic
MeSH Terms: conditions — Amyloidosis, Familial; Amyloid Neuropathies, Familial; Amyloid Neuropathies; Amyloidosis, Hereditary, Transthyretin-Related

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALN-TTRSC02 (Active Comparator)
  Interventions: Drug: ALN-TTRSC02
- Sterile normal saline 0.9% for SC administration (Placebo Comparator)
  Interventions: Drug: Sterile Normal Saline (0.9% NaCl)

INTERVENTIONS:
Drug: ALN-TTRSC02 — Ascending doses of ALN-TTRSC02 by subcutaneous (SC) injection
  Arms: ALN-TTRSC02
Drug: Sterile Normal Saline (0.9% NaCl) — Calculated volume to match active comparator
  Arms: Sterile normal saline 0.9% for SC administration

SUMMARY:
The purpose of this study is to determine the safety, tolerability, pharmacokinetics and pharmacodynamics of ALN-TTRSC02 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, age 18 to 65 years, inclusive.
* Body mass index (BMI) ≥18.0 kg/m2 and ≤30 kg/m2 assessed at Screening.
* No clinically significant health concerns, as determined by medical history and physical examination, in the opinion of the Investigator.
* Women of child bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be willing to use contraception, willing and able to comply with the study requirements and to provide written informed consent.
* For Japanese cohorts, subjects of Japanese descent are defined as people carrying a Japanese passport, descendants of 4 Japanese grandparents, and have not been outside Japan for more than 5 years.

Exclusion Criteria:

* Clinically relevant history or presence of respiratory, gastrointestinal, renal, cardiovascular, hepatic, hematological, lymphatic, neurological, psychiatric, musculoskeletal, genitourinary, immunological, and other inflammatory diseases, or dermatological or connective tissue diseases or disorders.
* Active serious mental illness or psychiatric disorder.
* Clinically significant ECG abnormalities. Abnormal for AST/ALT and any other clinical safety laboratory result considered clinically significant.
* Known history of allergic reaction to an oligonucleotide or GalNAc.
* History of intolerance to subcutaneous injection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-06-07 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2018-01-12 (Actual)

PRIMARY OUTCOMES:
Safety of ALN-TTRSC02, evaluated by the proportion of subjects experiencing adverse events (AEs) | Day 1 through to Day 314

SECONDARY OUTCOMES:
Profile of pharmacokinetics (PK) of ALN-TTRSC02 | Day 1 through to Day 3
  Cmax
Profile of pharmacokinetics (PK) of ALN-TTRSC02 | Day 1 through to Day 3
  tmax
Profile of pharmacokinetics (PK) of ALN-TTRSC02 | Day 1 through to Day 3
  AUC
Profile of pharmacokinetics (PK) of ALN-TTRSC02 | Day 1 through to Day 3
  t½
Profile of pharmacokinetics (PK) of ALN-TTRSC02 | Day 1 through to Day 3
  CL/F
Profile of pharmacokinetics (PK) of ALN-TTRSC02 | Day 1 through to Day 3
  Vss/F
Profile of pharmacokinetics (PK) of ALN-TTRSC02 | Day 1 through to Day 3
  Vz/F
Profile of pharmacokinetics (PK) of ALN-TTRSC02 | Day 1 through to Day 314
  fe
Profile of pharmacokinetics (PK) of ALN-TTRSC02 | Day 1 through to Day 314
  CLR
Effect of ALN-TTRSC02 on serum TTR levels as measured by reduction from baseline in serum TTR | Day 1 through to Day 314
Effect of ALN-TTRSC02 on serum Vitamin A levels as measured by reduction from baseline in serum Vitamin A | Screening through to Day 314

CONTACTS AND LOCATIONS:
Overall Officials: John Vest, MD, PhD, Study Director — Alnylam Pharmaceuticals
Locations (1):
- Clinical Trial Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Badri P, Kolachana K, Duong A, Lasko M, Nandi T, Mehrotra N, Robbie GJ. Platform Assessment of Concentration-QTc Relationship Across GalNAc-siRNA Molecules. Clin Pharmacokinet. 2025 Dec 12. doi: 10.1007/s40262-025-01606-0. Online ahead of print. PMID 41388232